CLINICAL TRIAL: NCT07033468
Title: The Feasibility and the Efficacy of the Full-immersive Virtual Reality Cognitive Training in Patients With Mild or Moderate Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202400517B0
Record Dates: First submitted 2025-03-25; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-02

CONDITIONS: Mild to Moderate Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR training therapy (Experimental): Guide the patient through a 5-minute warm-up, which mainly involves explaining, familiarizing with, or reviewing VR operations. After the warm-up, proceed with the first part of the VR gardening training for 10 minutes, followed by 5 minutes of eye and stretching exercises. Then, continue with the second part of the VR gardening training for another 10 minutes, followed by 5 minutes of eye massage and stretching exercises. This sequence is repeated for a total of four cycles.
  Interventions: Device: VR-WLC; Device: CTL-VR
- Waitlist control session (Other): During the waitlist period, patients will not receive any training but will receive regular phone calls to ensure equal attention.
  Interventions: Device: VR-WLC; Device: CTL-VR

INTERVENTIONS:
Device: VR-WLC — First, conduct the Virtual Reality (VR) training activity. After the evaluation is completed, proceed to the Waitlist Control (WLC) session, approximately 5 to 10 weeks later.
Device: CTL-VR — First, conduct the Control (CTL) session for approximately 5 to 10 weeks. After the evaluation is completed, proceed to the Virtual Reality (VR) training activity.

SUMMARY:
This project will explore the feasibility and efficacy of the fully immersive virtual reality leisure cognitive training tool developed by Chang Gung University in patients with mild to moderate dementia. The feasibility study will assess the feasibility and emotion-related indicators of 10 patients before and after a single training session. The efficacy study is planned to adopt a crossover randomized controlled trial, recruiting 30 patients for 15 sessions, each lasting 65 minutes, conducted three times a week. The assessment will include tests on the primary variable of cognitive function and secondary variables such as activities of daily living, quality of life, emotion, clinical symptoms, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 55 years;
2. Diagnosed with mild or moderate dementia (primarily degenerative dementia) by a consulting physician or based on past medical records;
3. A score of at least 11 but no more than 23 on the Mini-Mental State Examination (MMSE);
4. Has at least one family member or a regularly contacted friend (with the person's mobile number and contact at least once a week);
5. Able to walk independently and complete the Timed Up & Go (TUG) test;
6. Able to follow instructions with or without the assistance of a guardian or therapist;
7. If the assessment indicates moderate dementia, further evaluation will be conducted to determine whether the participant has sufficient capacity to provide informed consent. If their capacity is found to be impaired, the study will be explained to their legal representative

Exclusion Criteria:

1. Dementia with Lewy Bodies and other dementia types resulting from specific causes, such as Huntington's Disease, substance addiction, central nervous system infections, nutritional deficiencies, and metabolic disorders.
2. Severe health conditions that may hinder safe participation, such as respiratory distress, severe cardiovascular disease, or brain tumors.
3. A psychiatric diagnosis of psychosis within the past six months.
4. Diagnosis of Korsakoff syndrome.
5. History of substance addiction.
6. Severe hearing impairment or color blindness.
7. History of severe vertigo or epilepsy.
8. Concurrent participation in other studies that may affect cognitive function

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change scores of Montreal Cognitive Assessment | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  The Montreal Cognitive Assessment (MoCA) will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitive functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke.
  Minimum: 0 (worst performance) Maximum: 30 (best performance) The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Stroop test | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  The participants will be tested under congruent and incongruent conditions. In the congruent condition, the participant will name the color ink of a word which is consistent with the written color name; whereas in the incongruent condition the participant will name the color ink differs from the written color name. The time to complete the task will be calculated for each condition.Minimum: 0 , Maximum: but typically no upper limit. Higher scores indicate worse performance (greater cognitive interference and slower response time).
Change scores of Color trials test | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  For Part 1, the respondent uses a pencil to rapidly connect circles numbered 1-25 in sequence. For Part 2, the respondent rapidly connects numbered circles in sequence, but alternates between pink and yellow. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.Minimum: Greater than 1 second (best performance) Maximum: No upper limit .Higher scores indicate worse performance (longer completion time and greater cognitive impairment).
Change scores of Frontal Assessment Battery | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  This study utilizes this scale to assess various aspects of frontal lobe function, including executive function, behavioral regulation, and planning. The test consists of six subtests: Similarities, Verbal Fluency, Motor Sequencing, Conflicting Instructions, Go-No-Go, and Comprehending Behavior. Each subtest is scored from 0 to 3, with a total possible score of 18 points. The Taiwanese version of the frontal assessment scale has demonstrated good reliability and validity, showing consistency with tconsistency with the original version and strong construct validity.
  Minimum: 0 (worst performance) Maximum: 18 (best performance) Higher scores indicate better frontal lobe function, while lower scores suggest greater impairment.

SECONDARY OUTCOMES:
Change scores of Barthel Index | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  It is a commonly used assessment scale for evaluating activities of daily living (ADL), primarily designed to measure the effectiveness of treatment and the degree of functional decline in patients. The Barthel Index consists of 10 assessment items, each assigned a corresponding score (0, 5, or 10 points), with a maximum total score of 100 points. A lower total score indicates greater dependence on others and a reduced ability to perreduced ability to perform daily self-care activities.
Change scores of Amsterdam Instrumental Activity of Daily Living,A-IADL | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  The Amsterdam Instrumental Activity of Daily Living (A-IADL) is an adaptive and computerized questionnaire designed to assess impairments in instrumental activities of daily living (IADL) in (early) dementia. The questionnaire is completed by a caregiver, such as a relative or friend. Each item has a 5-point scale response option (scored 0-4). The scoring of the Amsterdam Instrumental Activity of Daily Living is calculated using item response theory .Lower scores indicating poorer performance. Higher scores indicate better performance in instrumental activities of daily living, while lower scores suggest greater impairment.
Change scores of The Chinese Dementia-Quality of Life instrument, DQoL | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  This study utilizes the Chinese version of the Quality of Life in Dementia (QOL-D) assessment tool to evaluate the physical and mental health of individuals with dementia and to understand the impact of VR cognitive training on their well-being. The questionnaire comprises five dimensions: positive emotions, negative emotions, sense of belonging, self-esteem, and aesthetics, with a total of 29 items. Each item is rated on a scale from 0 to 5, indicating varying levels of quality. This questionnaire is applicable to individuals with mild to moderate dementia, and its Chinese version has been validated among dementia patients in Taiwan.
  Minimum: 0 (worst quality of life) Maximum: 145 (best quality of life, calculated as 29 items × maximum score of 5 per item).
  Higher scores indicate better quality of life, while lower scores suggest poorer well-being.
Change scores of The Cornell Scale for Depression in Dementia Chinese version | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  This study utilizes the Chinese version of the Cornell Scale for Depression in Dementia (CSDD) to assess depressive symptoms in individuals with dementia before and after the intervention, aiming to understand the impact of the intervention on their quality of life. The scale covers five dimensions: mood-related signs, behavioral disturbances, physical signs, cyclic functions, and ideational disturbances, with a total of 19 items. Each item is scored based on severity, ranging from 0 (no symptoms) to 2 (severe symptoms). A total score above 10 suggests a possible diagnosis of depression, while a score below 6 indicates that depression can be ruled out. The Chinese version has established reliability and validity, demonstrating good psychometric properties.
  Minimum: 0 (no depressive symptoms) Maximum: 38 (severe depressive symptoms, calculated as 19 items × maximum score of 2 per item) Higher scores indicate more severe depressive symptoms, while lower scores suggest
Change scores of Clinical Dementia Rating, CDR | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  This study utilizes the Clinical Dementia Rating (CDR) scale to assess the severity of cognitive decline in individuals with dementia. The evaluation is conducted by professional physicians and clinical psychologists to comprehensively assess the cognitive function of participants. The assessment includes six functional domains: memory, orientation, judgment and problem-solving, community affairs, home and hobbies, and personal care. Based on the scoring criteria of the scale, a final score is derived to represent the current severity of dementia. This score serves as an important reference for tracking the progression of the disease over time. The Chinese version of the CDR scale has been validated and has demonstrated good reliability and validity Minimum: 0 (normal cognitive function) Maximum: 3 (severe dementia) Higher scores indicate more severe cognitive impairment.
Change scores of Behavioral and Psychological Symptoms of Dementia, BPSD | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  We use behavioral and psychological symptoms of dementia (BPSD) to assess the behavioral and psychological aspects of individuals with dementia. Dementia is not only characterized by cognitive impairment but is also frequently accompanied by non-cognitive symptoms such as depression, anxiety, delusions, hallucinations, behavioral disturbances, and other psychiatric symptoms. According to a past study conducted in Taiwan, the prevalence of non-cognitive symptoms among individuals with dementia was as high as 30% (Fuh & Liu, 2006). BPSD is also the primary source of burden for family caregivers of dementia patients. Additionally, compared to improvements in cognitive function, BPSD is often more noticeably improved in clinical settings.
  Minimum: 0 Maximum: Depends on the number of items and scoring system of the specific BPSD scale used Higher scores indicate more severe behavioral and psychological symptoms in individuals with dementia, while lower scores suggest fewer or no symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Tucheng Hospital, New Taipei City, commissioned and operated by Chang Gung Medical Foundation., New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided